CLINICAL TRIAL: NCT05978869
Title: The Effectiveness of Gamified Fitness Training Integrated Into Health Education to Promote Children's Physical Activity
Brief Title: Gamified Fitness Training to Promote Children's Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chi-Jane Wang (Other)
Responsible Party: Sponsor-Investigator, Chi-Jane Wang, Associate Professor, National Cheng-Kung University Hospital
Organization: National Cheng-Kung University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: A-ER-106-441
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Physical Activity Levels

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical fitness training (Experimental): The training group received physical fitness training for 12 weeks
  Interventions: Other: physical fitness training
- No training group (No Intervention): The no training group did not receive any training program

INTERVENTIONS:
Other: physical fitness training — Through a three-step process, gamified physical fitness training was developed by a multidisciplinary team.
  Arms: physical fitness training

SUMMARY:
The study aimed to introduce gamified physical fitness training in health education with the goal of enhancing physical activity levels and assessing its feasibility within a small-scale context involving 11-12-year-old children.

DETAILED DESCRIPTION:
A cluster experimental design was conducted in a small-scale context of school children. Participants were recruited by inviting two elementary schools located in the same district area for testing the physical fitness training effects. Two schools were randomly assigned to either the training group (TG; n = 47) receiving physical fitness training or the control group (CG; n = 44) without the training. Through a three-step process, gamified physical fitness training was developed by a multidisciplinary team from the TG school. PA outcome indicators were assessed using AI-wireless sensors attached to participants' wrists over 12 weeks. Participants' satisfaction was used to assess the feasibility of implementing gamified physical fitness training in health education classes. Data collection occurred during school days for one week at three-time points: the first week (T1), 6th week (T2), and the 12th week (T3). Generalized estimating equation statistics were used to assess the program effects.

ELIGIBILITY:
Inclusion Criteria:

* school children in 5th grade

Exclusion Criteria:

* physical deformity, mental disability, limited higher density physical activity such as asthma, cardiovascular disease, and bone fracture.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 91 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2018-12-15 (Actual)

PRIMARY OUTCOMES:
physical activity levels | week 0
  PA levels were measured in minutes spent on daily steps, total physical activity (TPA), light physical activity (LPA), moderate-to-vigorous physical activity (MVPA), and daily step counts using AI-wireless sensors attached to participants' wrists.
Learning Self-Efficacy | week 0
  Learning Self-Efficacy Scale (LSES) contains 18 items scored on a 5-point Likert scale with 4 items reversely scored. The total score of LSES ranges from -6 to 66, with higher scores reflecting higher LSE.
physical activity levels | week 6
  PA levels were measured in minutes spent on daily steps, total physical activity (TPA), light physical activity (LPA), moderate-to-vigorous physical activity (MVPA), and daily step counts using AI-wireless sensors attached to participants' wrists.
physical activity levels | week 12
  PA levels were measured in minutes spent on daily steps, total physical activity (TPA), light physical activity (LPA), moderate-to-vigorous physical activity (MVPA), and daily step counts using AI-wireless sensors attached to participants' wrists.
Learning Self-Efficacy | week 12
  Learning Self-Efficacy Scale (LSES) contains 18 items scored on a 5-point Likert scale with 4 items reversely scored. The total score of LSES ranges from -6 to 66, with higher scores reflecting higher LSE.

SECONDARY OUTCOMES:
Satisfaction levels | Week 12
  For the satisfaction of the PA program, the evaluation was conducted at the 12-week, encompassing five aspects: the integration of physical training into the HE classes, the content of the physical training, the application of gamification strategies in training, the active play during class breaks, and the effectiveness of GHPT in improving PA. Responses to levels of satisfaction with the training program were assessed across five categories: very satisfied, satisfied, OK, dissatisfied, and extremely dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Jane Wang, Ph.D., Principal Investigator — Department of Nursing, College of Medicine, National Cheng Kung University
Locations (1):
- Chi-Jane Wang, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No